CLINICAL TRIAL: NCT00952978
Title: Efficacy and Safety of Ilaprazole for Acute Duodenal Ulcer: A Randomized,Double-Blind,Omeprazole-Controlled,Multicenter,and Phase3 Trial in China
Brief Title: Ilaprazole for the Treatment of Duodenal Ulcer in Chinese Patients (Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Haitang Hu, Livzon Pharmaceutical Group Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Livzon-IY-81149-03; 2005L02943
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Duodenal Ulcer
Keywords: Ilaprazole; Proton pump inhibitor; Duodenal ulcer; Acid suppression; Randomized trial
MeSH Terms: conditions — Duodenal Ulcer | interventions — ilaprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mg ilaprazole (Experimental)
  Interventions: Drug: 10 mg ilaprazole
- 20 mg omeprazole (Active Comparator)
  Interventions: Drug: 20 mg omeprazole

INTERVENTIONS:
Drug: 10 mg ilaprazole — Two 5-mg ilaprazole tablets(Livzon Pharm Group Inc., China) together with one placebo capsule in a package being taken orally each morning on an empty stomach for 4 weeks
  Arms: 10 mg ilaprazole
Drug: 20 mg omeprazole — One 20-mg omeprazole capsule (AstraZeneca, Losec) together with two placebo tablets in a package being taken orally each morning on an empty stomach for 4 weeks
  Other Names: Losec,AstraZeneca
  Arms: 20 mg omeprazole

SUMMARY:
Patients with endoscopically diagnosed active duodenal ulcer disease were enrolled in a randomized, double-blind, parallel and positive-controlled trial. They were randomly assigned into two groups, 10 mg/day ilaprazole and 20 mg/day omeprazole, to be treated for up to four weeks and be seen at week 1, 2 and 4. The primary endpoint was the ulcer healing rate at week 4. Healing of ulcer was determined by its resolution from active to scarring stage. Symptoms relief was evaluated as secondary end points by using a graded score. Safety and tolerability were evaluated on basis of clinical assessments.

DETAILED DESCRIPTION:
The primary endpoint was the healing rate of ulcers, which based on post-treatment (week 4) endoscopic changes in stage of the ulcer relative to baseline (week 0) levels. Stages of the ulcers were endoscopically assessed according to the degree of ulceration, regenerating epithelialization, and scarring, which was defined as follows: A stage (active stage, A1 & A2) where A1 stage is more severe than A2 stage, H stage (healing stage, H1 & H2) where H2 stage is better than H1 stage, and S stage (scarring stage, S1 (red scar) & S2 (white scar)) where S stage is the best stage in the three stages and S2 stage is better than S1.Healing of ulcer is deemed successful if an ulcer in A stage resolved to S stage at the end of the treatment period, regardless of S1 or S2. When endoscopy demonstrated successful ulcer healing, study medication was discontinued. Patients returned at week 2, and if unhealed further endoscopic assessment would be done at week 4. Secondary endpoints included post-treatment resolution of related gastrointestinal symptoms such as upper abdominal pain, heartburn, acid regurgitation, nausea & vomiting, eructation, and increased flatus. These symptoms were recorded on a scale ranging from 0 to 3(0=none, 1=mild, 2=moderate, 3=severe) at baseline, week 1, 2, and 4. Resolution of symptoms were defined as "excellence", "effective", "improved", or "ineffective" relative to baseline levels, of which complete symptom relief or complete absence of the symptom without recurrence was deemed as "excellence". Safety assessments based mainly on the occurrence, frequency, and severity of adverse events, which were monitored throughout the duration of the study, and also based on comprehensive indexes, including physical examination, electrocardiography, and routine laboratory investigations, which were performed at baseline and repeated at the end of the treatment period. For all adverse events, where necessary, patients were withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients were eligible for enrollment if they:

  1. were 18-65 years of age,
  2. had endoscopically diagnosed active duodenal ulcers within the previous 72 hours and
  3. the number of ulcers was at least one, but no more than two with the larger diameter 0.3-2.0cm.

Exclusion Criteria:

* Patients were ineligible if they:

  1. had cancerous or complex ulcers, Zollinger-Ellison syndrome, esophageal erosion or ulcer, varices of esophagus or fundus of stomach, or pyloric stenosis,
  2. had a known history of gastric acid suppression operation, esophageal operation or peptic operation other than simple closure of perforation,
  3. had severe complications (e.g., pyloric obstruction, active bleeding under endoscope), severe other diseases of digestive tract such as Crohn's disease and ulcerative colitis, and severe other systemic diseases,
  4. were female patients who were breast feeding, pregnant, or intended to become pregnant during the study,
  5. had taken proton pump inhibitors within the 5 days or for more than three consecutive days within the two weeks immediately preceding start of study drug,
  6. participated in a clinical trial with an investigational drug or device within the past three months,
  7. had hypersensitivity or idiosyncratic reaction to omeprazole or any other benzimidazole,
  8. had alcoholic intemperance, drug addiction or any other improper habits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the healing rate of ulcers, which based on post-treatment (week 4) endoscopic changes in stage of the ulcer relative to baseline (week 0) levels. | week 4

SECONDARY OUTCOMES:
Secondary endpoints included post-treatment resolution of related gastrointestinal symptoms such as nightly pain, heartburn, nightly acid regurgitation, nausea & vomiting, eructation, and increased flatus. | week 4

CONTACTS AND LOCATIONS:
Overall Officials: S R Lin, M.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang L, Zhou L, Hu H, Lin S, Xia J. Ilaprazole for the treatment of duodenal ulcer: a randomized, double-blind and controlled phase III trial. Curr Med Res Opin. 2012 Jan;28(1):101-9. doi: 10.1185/03007995.2011.639353. Epub 2012 Jan 3. PMID 22070512